CLINICAL TRIAL: NCT04064320
Title: The Effect of Lullaby Intervention on Anxiety and Prenatal Attachment in Women With High-risk Pregnancy: A Randomised Controlled Study
Brief Title: The Effect of Lullaby Intervention on Anxiety and Attachment in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nazlı Baltacı, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 363
Record Dates: First submitted 2019-08-10; First posted 2019-08-21 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Anxiety; Attachment Disorder; Pregnancy Related
Keywords: pregnancy; high-risk; anxiety; prenatal attachment; bonding; lullaby; music
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Received lullaby intervention and usual care
  Interventions: Behavioral: Lullaby intervention
- Control group (No Intervention): No intervention other than usual care

INTERVENTIONS:
Behavioral: Lullaby intervention — Listening to lullabies, and accompanied by lullabies touching their abdomen and think about their babies of hospitalized women with high-risk pregnancy
  Arms: Intervention group

SUMMARY:
The aim of present study was to investigate the effect of lullaby intervention on anxiety and prenatal attachment in women with high-risk pregnancy. The study involved women with high-risk pregnancy who were assigned randomly to the intervention (n=30) or control (n=30) groups in a state hospital in Turkey. For two successive days, the intervention group listened to lullabies for 20 minutes once a day, meanwhile touched the abdomen and thought about their babies, but the control group did not. Data from the outcomes of anxiety and attachment were collected at baseline and at the end of the second day. Vital findings were measured on each study day, both before and after the lullaby intervention/usual care.

DETAILED DESCRIPTION:
Women with high-risk pregnancy may experience anxiety and low prenatal attachment due to many problems with pregnancy and hospitalization. It is reported that anxiety can have negative effects on prenatal attachment. The anxiety during pregnancy may adversely affect the health of the pregnant woman and fetus.

During the study period, 777 pregnant women were admitted to the clinic and 125 of them with high-risk pregnancy were assessed for eligibility for the study on 2 days a week. The pregnant women (n=76) who met the inclusion criteria and agreed to participate in the study were recruited. Participants were randomized in equal numbers to the intervention (n=38) and control groups (n=38) by withdrawing computer randomized sampling numbers (using Microsoft Excel 2010) from concealed envelopes to determine their group status. Participants were numbered according to their order of admittance to the hospital. After obtaining informed content and collecting baseline data, main researcher randomly chose one code for each woman. Data was collected together until the sample size was reached.

Participants were recruited by simple random sampling from the perinatology clinic at a state hospital in Turkey. An estimation of sample size was calculated at an effect size of 2.43 with a 5% level of significance on the primary outcome of anxiety in a sample study. According to G*power 3.1 31, each group required 30 participants. During the study, 125 women were assessed for eligibility, 49 of them were excluded. Some participants withdrew due to preterm birth (n=5), referral to another hospital (n=1) or discharged from hospital (n=10). Finally 60 participants who completed the lullaby intervention were included in data analysis. As a result of the study, the power of the test (α=0.05, 95% confidence interval) was 99.9% for each group n=30.

The preliminary study included five women at risk of preterm delivery who met the inclusion criteria. They were subjected to a lullaby intervention, and their study variables were evaluated. The women in the preliminary study were not included in the main study.

The IG listened to lullabies, and accompanied by lullabies touched their abdomen and thought about their babies. The CG received only the usual care of the hospital.

The lullaby recital consisted of 10 different lullabies with a mean duration of two minutes, for a total of 20 minutes.The lullabies were among the best-known ones from the Turkish culture. At the place of study, an academician of the Music Education Department of the University, Fine Arts Faculty was consulted regarding the lullaby recital.The pregnant women in the intervention group listened to the lullabies for 20 minutes per day, for two successive days using an MP3 player. To provide a homogeneous intervention and to avoid bias, the personal lullaby preferences of the pregnant women were ignored.

This intervention was performed in single patient rooms during bed rest, when the participants were available and felt ready. The doors and windows of the room was closed, and the participants were left alone. A disposable ear-tip was used for each participant. Before the initiation of the recital, the MP3 player was checked and the participants were instructed in the operation of the MP3 player (turning on, turning off, adjusting volume). The tempo of the lullaby was concordant with the normal heart rate (about 60-70 beats per minute), the participant determined and adjusted the volume to suit.

The control group received only the usual care of the hospital, resting in reclined position. All of the participants in both groups were ensured to have empty bladders and closed their cellphones, and none received any medical interventions during the lullaby intervention/usual care.

The study data was collected between 11:30 and 13:30 after lunch when no medical care, diagnostic tests or routine follow-up were administered. Initially, sociodemographic and obstetric data were collected by face-to-face interviews with participants. Intervention effect outcomes were anxiety and attachment which were measured at baseline. Anxiety was measured by the State-Trait Anxiety Inventory (STAI) and attachment was measured by the Prenatal Attachment Inventory (PAI). Before pregnant women filled the STAI and PAI, the instructions were read aloud to them and then they responded the questionnaires in silence. The STAI and PAI were reassessed at the end of the study (day 2) after the lullaby intervention/usual care. Vital findings were also measured on each study day, both before and after the lullaby intervention/usual care. The systolic and diastolic blood pressures and pulse rates of all participants were measured using a digital sphygmomanometer. The respiratory rate was measured by observing the chest and count the number of respirations out loud for one full minute using a digital watch while at bed rest (the same device was used for each participant). The level of satisfaction with listening to lullabies was assessed after the lullaby intervention at the end of the study using a 10-point Likert-type scale.

After the purposes and procedures of this study was explained, signed informed consent was obtained from all participants. Participants were assured of privacy and that their identity was protected. The study was based on voluntariness. Usual care and treatment of pregnant women in each groups were not intervened during the study period.

Data were analyzed by IBM SPSS v.23. Categorical data were analysed using the chi-square test for homogeneity of characteristics between two groups. Parametric tests were used if the data was normally distributed, but if not, nonparametric tests were used. A Pearson Chi-square test, Fisher's exact test, and Yates' continuity correction were used to compare the categorical data. The continuous data was compared using a Student's t or Mann-Whitney U-tests. A Paired sample t-test or Wilcoxon Signed Rank test were used to compare the paired scores of the STAI and PAI and the vital findings within the groups. The relationship between these three parameters was analyzed using a Spearman-correlation test. Statistical significance was considered p<0.05.

There are also some limitations in this study. Firstly, only state anxiety of the pregnant women was assessed, and future studies would benefit from taking also trait anxiety into consideration. It was a single-center study; therefore, the generalizability of the results to other women with high-risk pregnancy is unclear. Since the perinatology clinic where the study was carried out was newly opened, there were some disruptions and most pregnant women were transferred from this clinic to other clinics of hospital and discharged from hospital before the required hospital stay; therefore, the study could only be performed with pregnant women hospitalized for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization due to high-risk pregnancy
* 19 years and older
* Pregnancy duration longer than 28 weeks.
* Singleton pregnancy.
* Duration of hospitalization 24 hours minimum.
* Ability to read and write and to comprehend.
* Speaking Turkish.

Exclusion Criteria:

* Hospital admission due to severe preeclampsia, eclampsia or ablatio placenta.
* Presence of mental or cognitive disorders.
* Being under psychiatric treatment.
* Vision or hearing impairments.
* Fetal deformity or anomalies such as congenital diseases

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Anxiety change | At baseline and at the end of the 2nd day of study, anxiety was assessed.
  As assessed by the State-Trait Anxiety Inventory (STAI) STAI consists of two scales, a total of 40 self-reported items. The State Anxiety Scale only used in this study, consists of 20 straight and inverse scored terms, and is scored between 20 and 80 in a likert type scoring between 1 and 4. High scores indicate high anxiety levels.
Prenatal attachment change | At baseline and at the end of the 2nd day of study, prenatal attachment was assessed.
  As assessed by the Prenatal Attachment Inventory (PAI) PAI which is a likert type scale, has 21-item with four scores (1-4) and the total score is 21-84. A higher scores indicate higher levels of attachment.

SECONDARY OUTCOMES:
Change in Respiratory Rate | At 1st day of study before intervention/usual care, at 1st day of study after intervention/usual care, at 2nd day before intervention/usual care and at 2nd day after intervention/usual care
  The respiratory rate was measured by observing the chest and count the number of respirations out loud for one full minute using a digital watch while at bed rest. One respiration consists of one complete rise and fall of the chest (inhalation and exhalation of air).
Change in Heart Rate | At 1st day of study before intervention/usual care, at 1st day of study after intervention/usual care, at 2nd day before intervention/usual care and at 2nd day after intervention/usual care
  The heart rate was measured using a digital sphygmomanometer.
Change in Systolic Blood Pressure | At 1st day of study before intervention/usual care, at 1st day of study after intervention/usual care, at 2nd day before intervention/usual care and at 2nd day after intervention/usual care
  The systolic blood pressure was measured using a digital sphygmomanometer and recorded in mmHg.
Change in Diastolic Blood Pressure | At 1st day of study before intervention/usual care, at 1st day of study after intervention/usual care, at 2nd day before intervention/usual care and at 2nd day after intervention/usual care
  The diastolic blood pressure was measured using a digital sphygmomanometer and recorded in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Baltacı, phD, Principal Investigator — Ondokuz Mayıs University, Assistant Professor phD; Mürüvvet Başer, Professor, Study Director — Erciyes University, Professor
Locations (1):
- Ondokuz Mayıs University, Faculty of Health Sciences, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arabin B, Jahn M. "Need for interventional studies on the impact of music in the perinatal period: results of a pilot study on women's preferences and review of the literature". J Matern Fetal Neonatal Med. 2013 Mar;26(4):357-62. doi: 10.3109/14767058.2012.733763. Epub 2012 Nov 1. PMID 23039049
- [Background] Bauer CL, Victorson D, Rosenbloom S, Barocas J, Silver RK. Alleviating distress during antepartum hospitalization: a randomized controlled trial of music and recreation therapy. J Womens Health (Larchmt). 2010 Mar;19(3):523-31. doi: 10.1089/jwh.2008.1344. PMID 20141383
- [Background] Arranz Betegon A, Garcia M, Pares S, Montenegro G, Feixas G, Padilla N, Camacho A, Goberna J, Botet F, Gratacos E. A Program Aimed at Reducing Anxiety in Pregnant Women Diagnosed With a Small-for-Gestational-Age Fetus: Evaluative Findings From a Spanish Study. J Perinat Neonatal Nurs. 2017 Jul/Sep;31(3):225-235. doi: 10.1097/JPN.0000000000000270. PMID 28737543
- [Background] Carolan-Olah M, Barry M. Antenatal stress: an Irish case study. Midwifery. 2014 Mar;30(3):310-6. doi: 10.1016/j.midw.2013.03.014. Epub 2013 May 16. PMID 23684696
- [Background] Carolan M, Barry M, Gamble M, Turner K, Mascarenas O. The Limerick Lullaby project: an intervention to relieve prenatal stress. Midwifery. 2012 Apr;28(2):173-80. doi: 10.1016/j.midw.2010.12.006. Epub 2011 Mar 3. PMID 21371795
- [Background] Carolan M, Barry M, Gamble M, Turner K, Mascarenas O. Experiences of pregnant women attending a lullaby programme in Limerick, Ireland: a qualitative study. Midwifery. 2012 Jun;28(3):321-8. doi: 10.1016/j.midw.2011.04.009. Epub 2011 Jun 8. PMID 21641704
- [Background] Chang MY, Chen CH, Huang KF. Effects of music therapy on psychological health of women during pregnancy. J Clin Nurs. 2008 Oct;17(19):2580-7. doi: 10.1111/j.1365-2702.2007.02064.x. Epub 2008 Feb 19. PMID 18298503
- [Background] Chang HC, Yu CH, Chen SY, Chen CH. The effects of music listening on psychosocial stress and maternal-fetal attachment during pregnancy. Complement Ther Med. 2015 Aug;23(4):509-15. doi: 10.1016/j.ctim.2015.05.002. Epub 2015 May 27. PMID 26275644
- [Background] Corbijn van Willenswaard K, Lynn F, McNeill J, McQueen K, Dennis CL, Lobel M, Alderdice F. Music interventions to reduce stress and anxiety in pregnancy: a systematic review and meta-analysis. BMC Psychiatry. 2017 Jul 27;17(1):271. doi: 10.1186/s12888-017-1432-x. PMID 28750631
- [Background] Ding XX, Wu YL, Xu SJ, Zhu RP, Jia XM, Zhang SF, Huang K, Zhu P, Hao JH, Tao FB. Maternal anxiety during pregnancy and adverse birth outcomes: a systematic review and meta-analysis of prospective cohort studies. J Affect Disord. 2014 Apr;159:103-10. doi: 10.1016/j.jad.2014.02.027. Epub 2014 Feb 26. PMID 24679397
- [Background] Dipietro JA. Psychological and psychophysiological considerations regarding the maternal-fetal relationship. Infant Child Dev. 2010;19(1):27-38. doi: 10.1002/icd.651. PMID 20228872
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Garcia Gonzalez J, Ventura Miranda MI, Manchon Garcia F, Pallares Ruiz TI, Marin Gascon ML, Requena Mullor M, Alarcon Rodriguez R, Parron Carreno T. Effects of prenatal music stimulation on fetal cardiac state, newborn anthropometric measurements and vital signs of pregnant women: A randomized controlled trial. Complement Ther Clin Pract. 2017 May;27:61-67. doi: 10.1016/j.ctcp.2017.03.004. Epub 2017 Apr 1. PMID 28438283
- [Background] Garcia-Gonzalez J, Ventura-Miranda MI, Requena-Mullor M, Parron-Carreno T, Alarcon-Rodriguez R. State-trait anxiety levels during pregnancy and foetal parameters following intervention with music therapy. J Affect Disord. 2018 May;232:17-22. doi: 10.1016/j.jad.2018.02.008. Epub 2018 Feb 13. PMID 29471206
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Background] Littleton HL, Breitkopf CR, Berenson AB. Correlates of anxiety symptoms during pregnancy and association with perinatal outcomes: a meta-analysis. Am J Obstet Gynecol. 2007 May;196(5):424-32. doi: 10.1016/j.ajog.2007.03.042. PMID 17466693
- [Background] Liu YH, Lee CS, Yu CH, Chen CH. Effects of music listening on stress, anxiety, and sleep quality for sleep-disturbed pregnant women. Women Health. 2016;56(3):296-311. doi: 10.1080/03630242.2015.1088116. Epub 2015 Sep 11. PMID 26361642
- [Background] Muller ME. Development of the Prenatal Attachment Inventory. West J Nurs Res. 1993 Apr;15(2):199-211; discussion 211-5. doi: 10.1177/019394599301500205. No abstract available. PMID 8470375
- [Background] Ossa X, Bustos L, Fernandez L. Prenatal attachment and associated factors during the third trimester of pregnancy in Temuco, Chile. Midwifery. 2012 Oct;28(5):e689-96. doi: 10.1016/j.midw.2011.08.015. Epub 2011 Sep 28. PMID 21955858
- [Background] Persico G, Antolini L, Vergani P, Costantini W, Nardi MT, Bellotti L. Maternal singing of lullabies during pregnancy and after birth: Effects on mother-infant bonding and on newborns' behaviour. Concurrent Cohort Study. Women Birth. 2017 Aug;30(4):e214-e220. doi: 10.1016/j.wombi.2017.01.007. Epub 2017 Feb 4. PMID 28169158
- [Background] Pisoni C, Garofoli F, Tzialla C, Orcesi S, Spinillo A, Politi P, Balottin U, Manzoni P, Stronati M. Risk and protective factors in maternal-fetal attachment development. Early Hum Dev. 2014 Sep;90 Suppl 2:S45-6. doi: 10.1016/S0378-3782(14)50012-6. PMID 25220127
- [Background] Shin HS, Kim JH. Music Therapy on Anxiety, Stress and Maternal-fetal Attachment in Pregnant Women During Transvaginal Ultrasound. Asian Nurs Res (Korean Soc Nurs Sci). 2011 Mar;5(1):19-27. doi: 10.1016/S1976-1317(11)60010-8. Epub 2011 Apr 5. PMID 25029946
- [Background] Toker E, Komurcu N. Effect of Turkish classical music on prenatal anxiety and satisfaction: A randomized controlled trial in pregnant women with pre-eclampsia. Complement Ther Med. 2017 Feb;30:1-9. doi: 10.1016/j.ctim.2016.11.005. Epub 2016 Nov 18. PMID 28137517
- [Background] Yang M, Li L, Zhu H, Alexander IM, Liu S, Zhou W, Ren X. Music therapy to relieve anxiety in pregnant women on bedrest: a randomized, controlled trial. MCN Am J Matern Child Nurs. 2009 Sep-Oct;34(5):316-23. doi: 10.1097/01.NMC.0000360425.52228.95. PMID 19713801